CLINICAL TRIAL: NCT07263945
Title: Influence of Prosthetic Foot Stiffness on Transtibial Osseointegrated Bone-Anchored Limb Outcomes
Acronym: TBAL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 25-0854; 1R01HD119003-01 (NIH)
Record Dates: First submitted 2025-10-22; First posted 2025-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Amputation; Transtibial Amputation - Unilateral; Bone Anchored Devices; Osseointegration
Keywords: amputation; bone anchored limb; osseointegration; transtibial amputation; below knee amputation; prosthetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two prosthetic foot stiffness categories stiffer than the as-prescribed prosthetic foot stiffness (Active Comparator): A prosthetic foot that is two prosthetic foot stiffness categories stiffer than the stiffness of the as-prescribed prosthetic foot. The prosthetic foot type, including the manufacturer and length, will remain the same as the nominal (as-currently prescribed) foot.
  Interventions: Device: A prosthetic foot that is two prosthetic foot stiffness categories softer than the stiffness of the as-prescribed prosthetic foot
- Two prosthetic foot stiffness categories softer than the as-prescribed prosthetic foot stiffness (Active Comparator): A prosthetic foot that is two prosthetic foot stiffness categories softer than the stiffness of the as-prescribed prosthetic foot. The prosthetic foot type, including the manufacturer and length, will remain the same as the nominal foot.
  Interventions: Device: A prosthetic foot that is two prosthetic foot stiffness categories stiffer than the stiffness of the as-prescribed prosthetic foot
- As-prescribed prosthetic foot stiffness (Active Comparator): The prosthetic foot that is currently prescribed and used by each participant daily.
  Interventions: Device: As-prescribed prosthetic foot stiffness

INTERVENTIONS:
Device: As-prescribed prosthetic foot stiffness — Each participant will complete a motion capture collection, tests of physical function, and sensory tests in their currently prescribed prosthetic foot.
  Arms: As-prescribed prosthetic foot stiffness
Device: A prosthetic foot that is two prosthetic foot stiffness categories stiffer than the stiffness of the as-prescribed prosthetic foot — Each participant will complete a motion capture collection, tests of physical function, and sensory tests in a prosthetic foot that is two categories stiffer than their currently prescribed prosthetic foot.
  Arms: Two prosthetic foot stiffness categories softer than the as-prescribed prosthetic foot stiffness
Device: A prosthetic foot that is two prosthetic foot stiffness categories softer than the stiffness of the as-prescribed prosthetic foot — Each participant will complete a motion capture collection, tests of physical function, and sensory tests in a prosthetic foot that is two categories softer than their currently prescribed prosthetic foot.
  Arms: Two prosthetic foot stiffness categories stiffer than the as-prescribed prosthetic foot stiffness

SUMMARY:
A clinical trial utilizing cross-over study design in which individuals with transtibial amputation using either a bone-anchored limb or standard socket prosthesis will perform activities of daily living with varying prosthetic foot stiffness categories to complete the following 4 Specific Aims: 1) Determine the influence of prosthetic foot stiffness on dynamic bone-implant loading, 2) Determine how prosthetic foot stiffness influences function, pain, and multi-joint biomechanics outcomes, 3) Establish how prosthetic foot stiffness influences osseoperception and fall risk, and 4) Establish target ranges of optimal foot stiffness based on the sensitivity biomechanical outcomes to variability in foot stiffness.

DETAILED DESCRIPTION:
This will be a clinical trial with two groups (individuals with a unilateral transtibial amputation using either an osseointegrated bone-anchored limb or socket prosthesis that will implement a cross-over design. The objective of this clinical trial is to determine how changes in prosthetic foot stiffness influence clinical and biomechanical outcomes in patients with transtibial osseointegrated bone-anchored limbs compared to patients with transtibial amputation using a standard socket-suspended prosthesis. Although proper loading between the bone and implant is pivotal to promote and maintain osseointegration, which is required for physiological loading and thus positive outcomes, evidence surrounding the role of how prosthetic componentry influences force transmission and functional outcomes in this population currently does not exist. The findings of this clinical trial will address a critical knowledge gap pertaining to the role of componentry on multi-loading domain outcomes. Outcomes will be assessed in each participant in the same three conditions: one with their clinical prescribed prosthetic foot, one with a soft prosthetic foot (-2 stiffness categories less than prescribed), and one with a stiff prosthetic foot (+2 stiffness categories more than prescribed). This data will be used to test/develop the following aims: 1) Does foot stiffness change loading between the bone and implant during activities of daily living? 2) Does foot stiffness influence measures of function, pain, and biomechanics in patients with transtibial osseointegrated bone-anchored limbs differently than a socket prosthesis? 3) Does foot stiffness influence sensitivity, balance, and fall risk in patients using an osseointegrated bone-anchored limb different than a socket prosthesis? and 4) (exploratory) develop an optimization platform using computer models to determine the optimal foot stiffness that maximizes joint loading symmetry and minimizes metabolic cost.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation due to traumatic, congenital, or cancer-related causes
* > 12-months bone-anchored limb implantation surgery (Bone Anchored Limb group)
* > 12-months limb amputation (Socket Control group)
* Non-vascular amputation etiology
* Low profile prosthetic foot (nominal)
* Can walk unassisted for 5-minutes
* > 18 years old

Exclusion Criteria:

* Major amputation on contralateral limb
* Vascular amputation etiology
* Neurologic pathology that impairs coordination/balance
* Regular assistive device use required for community ambulation
* Inflammatory diseases or diabetes
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Bone-Implant Stress/Strain Impulse during Decline Walking (internal) | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Stress/strain impulse at the bone-implant interface (area under time series curve) will be calculated during the stance period of the decline walk (-5 degrees). Subject-specific finite element models will be developed for each bone-anchored limb participant to calculate this outcome. This will be done by including each participant's movement patterns, muscle forces, joint forces, bone geometry and bone health. Movement patterns, muscle forces, and joint loading will be calculated from musculoskeletal modeling using whole-body motion data collected from 70 wearable reflective markers (Vicon, Centennial, CO), ground reaction forces simultaneously collected from an instrumented treadmill (Bertec, Columbus, OH). Bone geometry and healthy will be determined from quantitative computed tomography bone scans.

SECONDARY OUTCOMES:
Bone-Implant Dynamic Stress/Strain Impulse (internal) | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Stress/strain impulse at the bone-implant interface (area under time series curve) will be calculated for each bone-anchored limb participant using motion and force data collected during the stance period of treadmill walking at level and incline (+5 degree) angles.
Bone Dynamic Stress/Strain Impulse (internal) | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Stress/strain impulse for the amputated tibia bone (area under time series curve) will be calculated for each bone-anchored limb participant using motion and force data collected during the stance period of treadmill walking at level, incline (+5 degree), and decline (-5 degree) angles.
Implant Dynamic Stress/Strain Impulse (internal) | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Stress impulse for the prosthesis implant (area under time series curve) will be calculated for each bone-anchored limb participant using motion and force data collected during the stance period of treadmill walking at level, incline (+5 degree), and decline (-5 degree) angles.
Prosthesis Force Impulse (external abutment) | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Force impulse in the vertical direction (area under the time series curve) will be calculated for all study participants using motion and force data collected from the triaxial load sensor in the prosthesis (iPECSTM) during the stance period of treadmill walking at level, incline (+5 degree), and decline (-5 degree) angles.
Sensory Threshold | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  With each foot (stiff, nominal (as-prescribed), soft), participants will stand on a platform with the prosthetic equivalent of the head of the third metatarsal in contact with an extension pin delivering a vibration. While wearing noise-reducing headphones, three different vibration frequencies will be tested in a randomized order: 8, 32, and 125 Hz. At each frequency, custom software will increase and decrease the vibrational amplitude at a rate of 0.2 dB/s. Using an integrated push button, the participant will indicate when sensation is felt (during increasing amplitude) or when sensation is lost (during decreasing amplitude), which will be the sensory threshold.
Postural Sway | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Postural sway will be quantified during quiet standing with eyes open and eyes closed condition. Using the center of pressure measured from the force platform under both feet, path length and 95% confidence ellipse area will be calculated.
Reactive Postural Control Time | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Reaction times during stepping responses to rapid treadmill belt perturbations will be measured using a force-instrumented treadmill (Bertec, Columbus, OH, USA).
Whole-Body Angular Momentum | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Peak-to-peak whole-body angular momentum will be calculated as a measure of dynamic balance during each dynamic functional activity (level/incline/decline walking and stair ascent/descent) and treadmill perturbation.
Self-Selected Gait Speed | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Gait velocity will be calculated using the time it takes each participant to walk 5-meters at their preferred, self-selected pace, averaged over three trials.
L-Test Time | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  The L-test will be quantified as the time it takes to stand up from a chair, walk 3-meters, complete a 90° left turn, walk 7-meters, completed a 180° turn, walk back on the same path, turn, and sit down.
Acceptability of Intervention Measure | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  The Acceptability of Intervention Measure is a 4-item, Likert-scale (5 point) self-report questionnaire assessing participant acceptability of the intervention (prosthetic foot type). Final scores range from 1 to 5 points, as the mean of the four items, with higher scores indicating greater acceptability.
Prosthetic Limb Users Survey of Mobility | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  The Prosthetic Limb Users Survey of Mobility is a 12-item, Likert scale (5 point) self-report questionnaire assessing participant mobility when using a prosthesis. Final scores range from 12 to 60 points with higher scores indicating greater mobility.
Activities-Specific Balance Confidence Scale | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  The Activities-Specific Balance Confidence Scale is a 16-item, 0-100 scale, self-reported questionnaire assessing participant balance confidence. Final scores range from 0% (no confidence in balance) to 100% (complete confidence in balance).
Joint Reaction Force | Three laboratory visits, each lasting approximately 4 hours, spanning across approximately 6-8 weeks
  Bilateral hip and knee joint reaction forces (normalized to body weight) will be calculated during treadmill walking using a combination of motion-capture data and subject-specific musculoskeletal models.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish the trial results data on the ClinicalTrials.gov website, on which the clinical trial will be registered. Sharing of data will include the potential of sharing raw data generated from all clinical assessments under a data-sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: The investigators will publish the trial results within one year of testing the final participant.
Access Criteria: User registration will be required to access/download any data and will require agreement to conditions of use in accordance with CDMRP Policy on Sharing Data and Research Resources.